CLINICAL TRIAL: NCT00801125
Title: A Phase IV, Open-Label Study of Tysabri (Natalizumab) in Patients Who Failed Anti-TNF-α Therapy
Brief Title: Study of Tysabri (Natalizumab) in Patients Who Failed Anti-TNF-α Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study sponsor decided to withdraw the current study prior to enrollment of first participant.
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELN51-309-503; CD FACTOR
Record Dates: First submitted 2008-12-01; First posted 2008-12-03 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2009-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Natalizumab

INTERVENTIONS:
Drug: natalizumab
  Other Names: TYSABRI

SUMMARY:
The purpose of this study is to demonstrate the safety, tolerability and clinical benefit of TYSABRI® (natalizumab) in patients with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be able and willing to give written informed consent and to comply with the requirements of this study protocol;
2. All patients must be CD TOUCH™ Prescribing Program enrolled;
3. Male or female patients, ≥ 18 years of age;
4. Patients with at least a 3-month history of CD;
5. Patients with clinical evidence of active (symptomatic) CD based on clinical history and radiologic or endoscopic findings within the previous 36 months. Patients with active disease following surgical resection must have radiological or endoscopic confirmation of CD post-surgery;
6. Patients must have evidence of active inflammation measured by CRP >2.87mg/L at the Screening visit;
7. Subjects must have a CDAI score ≥ 220 and ≤ 450 at Week 0;
8. Female patients must utilize a highly effective method of birth control throughout the study and for 3 months after study completion, or female patients must not be of childbearing potential, defined as postmenopausal at least two years, or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy);
9. Initial treatment with an approved anti-TNF-α therapy, specifically infliximab, adalimumab, or certolizumab, who had either a primary or secondary treatment failure, or intolerance, to those agents;

   1. A primary treatment failure is defined as one of the following:

      * The minimal requirement for a primary treatment failure to infliximab is defined as failure to respond to an induction regimen of 5 mg/kg at weeks 0, 2, and 6;
      * The minimal requirement for a primary treatment failure to adalimumab is defined as failure to respond to an induction regimen of 160 mg at week 0, and 80 mg at week 2;
      * The minimal requirement for a primary treatment failure to certolizumab is defined as a failure to respond to an induction regimen of 400 mg at weeks 0, 2, and 4;
   2. Secondary failures to a single anti-TNF-α agent is defined as:

      * experienced clinical benefit in the opinion of the investigator, but lost that benefit over time or discontinued due to an adverse event, and / or;
      * experienced clinical benefit in the opinion of the investigator, but are unable to be discontinued from concurrent oral corticosteroid therapy (i.e. ≥ 10 mg/day of prednisone/prednisolone or equivalent).
   3. Secondary failures to two anti-TNF-α agents is defined as:

      * experienced clinical benefit to their initial anti-TNF-α agent in the opinion of the investigator, lost that benefit over time or discontinued due to an adverse event, and failed to regain clinical benefit following the administration of a standard induction protocol to a second anti-TNF-α agent; and/or;
      * experienced clinical benefit in the opinion of the investigator, but are unable to be discontinued from concurrent oral corticosteroid therapy (i.e. ≥ 10 mg/day of prednisone/prednisolone or equivalent).
10. Intolerance is defined as an inability to tolerate additional administration of an agent due to acute or delayed reactions, as defined by the investigator;
11. Adequate cardiac, renal and hepatic function as determined by principal investigator and demonstrated by screening laboratory evaluations, questionnaires, and physical examination results that are within normal limits.

Exclusion Criteria:

1. Women of childbearing potential unless surgically sterile or using adequate contraception (IUD, oral or depot contraceptive, or barrier plus spermicide), and willing and able to continue contraception for 3 months after the last infusion of study drug (i.e., up to Week 20). Women using oral contraception must have started using it at least 2 months prior to enrollment;
2. Women who are pregnant or breastfeeding;
3. Prior treatment with TYSABRI® (natalizumab) (also referred to as Antegren™ in previous clinical trials);
4. Symptoms suggestive of intestinal stricture or obstruction;
5. History of cancer or lymphoproliferative disease other than a successfully and completely treated squamous cell or basal cell carcinoma of the skin;
6. Patients with a history of Listeria or human immunodeficiency virus (HIV) or a history of previously untreated TB;
7. Patients who have had surgical bowel resections in the past 2 weeks or are planning any resection within 4 weeks of starting the study medication;
8. Patients who do not meet any of the following criteria regarding baseline medications for CD (Please note that the term "Week 0" below refers to the exact day of the baseline visit):

   1. Baseline use of anti-tumor necrosis factor (anti-TNF-α) therapy, or previous use of all three approved agents, is not permitted;
   2. Baseline use of azathioprine (AZA), 6 mercaptopurine (6MP) / 6 thioguanine (6TG) / methotrexate (MTX) is not permitted;
   3. Baseline use of any other immunosuppressant (e.g., tacrolimus, cyclosporin, mycophenolate mofetil or leflunomide) is not permitted;
   4. Experimental agents must have been discontinued at least 4 weeks prior to Week 0, or for a period equivalent to 5 half-lives (t½) of the agent (whichever is longer);
   5. Any baseline 5-Aminosalicylate (5 ASA) compounds or antibiotics are permitted and if used must be continued at a stable dose during the trial;
   6. Any baseline 5-Aminosalicylate (5 ASA) compounds or antibiotics must have been administered at a stable dose for a minimum of 4 weeks prior to Week 0;
   7. Any baseline use of budesonide must have been administered at a stable dose for a minimum of 2 weeks prior to Week 0;
   8. For oral steroids other than budesonide, patients must have been at a stable dose for a minimum of 2 weeks prior to Week 0;
9. Patients likely to require emergency surgery for persistent intestinal obstruction, bowel perforation, uncontrolled bleeding or abdominal abscess infection, and patients who have undergone bowel surgery, including resections, within the 3 months prior to Week 0;
10. Patients who have a colostomy, ileostomy, or colectomy with ileorectal anastomosis;
11. Ileal resections resulting in clinically relevant short bowel syndrome, in the opinion of the Investigator;
12. Patients who are receiving or have received nasogastric/nasoenteric tube feeding, an elemental diet, or total parenteral nutrition (TPN) within the 2 weeks prior to Week 0;
13. Patients with a chest X-ray suggestive of pulmonary infection at screening;
14. Patients with a history of clinically significant and/or persistent gastrointestinal disorder (other than CD), cardiovascular, renal, hepatic, neurological, dermatological, immunological, major psychiatric (including drug or alcohol abusers), or hematological illness;
15. Patients with any laboratory tests considered clinically significant at screening;
16. Patients whose symptoms are likely caused by factors other than inflammatory CD, including infection, irritable bowel syndrome (IBS), or ulcerative colitis (UC);
17. Patients who will be unavailable for the duration of the trial, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason;
18. Patients who have do not have evidence of active inflammation.
19. Patients with active opportunistic infection or history of opportunistic infection in the last 6 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) achieving a clinical response at Week 12, defined as a reduction in the CDAI score from baseline (Week 0) of ≥ 70 points.

SECONDARY OUTCOMES:
Proportion (%) achieving a clinical remission at each visit, defined as a CDAI score < 150
Proportion achieving clinical response at Week 4 and Week 8
Proportion achieving a ≥ 100 point decrease in baseline (Week 0) CDAI score at each visit